CLINICAL TRIAL: NCT04587986
Title: Efficacy of Simultaneous Application of Noninvasive Repetitive Pulse Magnetic Stimulation (rPMS) and Radiofrequency for Abdominal Toning and Reduction of Subcutaneous Fat: Single-Blind Randomized Sham-Controlled Trial
Brief Title: rPMS and Radiofrequency for Abdominal Toning and Reduction of Subcutaneous Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTL-703_200
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Fat Burn

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Abdominal Toning and Reduction of Subcutaneous Fat (Experimental): The treatment administration phase will consist of three (3) treatments, delivered once a week. The applicator of BTL-703 will be applied over the umbilicus. The active group will receive treatment with intensities of a magnetic field and radiofrequency energy just below the patient's tolerance threshold. The device will induce visible muscle contractions along with heating of the subcutaneous fat.
  Interventions: Device: BTL-899
- Sham control (Sham Comparator): The treatment administration phase will also consist of three (3) treatments, delivered once a week. The sham group will receive a treatment with the intensities of the magnetic field and radiofrequency energy set to 5% of the maximum device output.
  Interventions: Device: BTL-899

INTERVENTIONS:
Device: BTL-899 — Treatment with intensities of a magnetic field and radiofrequency energy just below the patient's tolerance threshold.

SUMMARY:
This study will evaluate the clinical efficacy and safety of a simultaneous treatment by high power magnet and radiofrequency energy for toning of abdomen and reduction of subcutaneous fat. The study is a prospective multi-center single-blinded sham-controlled study. The subjects will be enrolled and assigned into two study groups; active and sham group. Subjects of both groups will be required to complete three (3) treatment visits and two to three follow-up visits.

DETAILED DESCRIPTION:
This study will evaluate the clinical efficacy and safety of a simultaneous treatment by high power magnet and radiofrequency energy for toning of abdomen and reduction of subcutaneous fat. The study is a prospective multi-center single-blinded sham-controlled study. The subjects will be enrolled and assigned into two study groups; active and sham group. Subjects of both groups will be required to complete three (3) treatment visits and two to three follow-up visits.

At the baseline visit, ultrasound imaging will be performed; the subject's weight and waist circumference will be recorded. Photos of the treated area will be taken.

The treatment administration phase in both study groups will consist of three (3) treatments, delivered once a week. The applicator of BTL-703 will be applied over the umbilicus. The active group will receive treatment with intensities of a magnetic field and radiofrequency energy just below the patient's tolerance threshold. The device will induce visible muscle contractions along with heating of the subcutaneous fat. The sham group will receive a treatment with the intensities of the magnetic field and radiofrequency energy set to 5% of the maximum device output.

At the last therapy visit, the subject's weight and waist circumference will be recorded, and photos of the treated area will be taken. In addition, subjects will receive Subject Satisfaction Questionnaire to fill in.

Safety measures will include documentation of adverse events (AE) including the subject's experience of pain or discomfort after each procedure. Following each treatment administration and at all of the follow-up visits, subjects will be checked for immediate post-procedure adverse event assessment.

During the post-procedure visits (at 1-month and 3-month follow-up visits), the subjects will undergo ultrasound imaging. Also, the subject's satisfaction will be noted, and weight with waist circumference will be recorded. Photographs of the treated area will be taken. There will be an option of a 6-months follow-up visit, according to subject's availability.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent form
* BMI ≤ 35 kg/m2
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring during study participation
* Subjects willing and able to maintain her regular (pre-procedure) diet and exercise regimen without affecting significant change in either direction during study participation

Exclusion Criteria:

* Electronic implants (such as cardiac pacemakers, defibrillators, and neurostimulators)
* Metal implants
* Drug pumps
* Malignant tumor
* Pulmonary insufficiency
* Injured or otherwise impaired muscles
* Cardiovascular diseases
* Disturbance of temperature or pain perception
* Hemorrhagic conditions
* Septic conditions and empyema
* Acute inflammations
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contagious skin disease
* Elevated body temperature
* Pregnancy, postpartum period, nursing, and menstruation
* Intrauterine device (IUD)
* Swollen or neoplastic tissues, space-occupying lesions or skin eruptions in the treatment area
* Basedow's disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Changes in fat and muscle thickness in the abdominal area measured via ultrasound. | 7 months
  To gather clinical evidence on the effectiveness of the combined treatment for abdominal toning and subcutaneous fat reduction through changes in abdominal tissues, measured via ultrasound and comparison of active and sham groups. The changes will be considered statistically significant where p-value <0.05.

SECONDARY OUTCOMES:
Patient's satisfaction with study treatment measured via questionnaires | 7 months
  To determine the patient's satisfaction with study treatment for non-invasive aesthetic improvement of the abdomen. The 5-point Likert scale Satisfaction questionnaire will be used to evaluate the participant's satisfaction with the therapy outcome. Subject satisfaction will be assessed after the last therapy visit and during the follow-up visits.
Evaluation of the Therapy's Safety Measured Via Therapy Comfort Questionnaire | 7 months
  The outcome will further be measured through the occurrence of adverse events or lack thereof. On Numerical Analog Scale (0-10), where 0 represents 'no pain' and 10 represents 'worst possible pain' select the level of pain experienced during the treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Julene B. Samuels, River Bluff, Kentucky
  - Maryland Laser Skin and Vein Institute, Hunt Valley, Maryland
  - JUVA Skin & Laser Center, New York, New York

IPD SHARING:
Plan to Share IPD: No